CLINICAL TRIAL: NCT02168634
Title: The Use of Botulinum Toxin in the Treatment of Itching From Hypertrophic Scar -- A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Kuei-Chang Hsu, Attending Physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGHKS13-CT12-23
Record Dates: First submitted 2014-03-11; First posted 2014-06-20 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Itchiness; Hypertrophic Scar; Botulinum Toxin
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Botulinum toxin (Experimental): 5U Botulinum toxin in 1cc normal saline, administered in one of the two itchy points
  Interventions: Drug: Botulinum Toxins
- Normal Saline (Placebo Comparator): 1cc normal saline, administered in the other itchy point
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxins — 5U botulinum toxin in 1c.c. normal saline, local injection
  Arms: Botulinum toxin
Drug: Placebo — 1cc normal saline, local injection
  Arms: Normal Saline

SUMMARY:
Hypertrophic scar, a disfiguring tissue reaction to trauma, occurred in around 20 % of the population. The patients with hypertrophic scar usually seek medical assistance not just for the annoying appearance but mostly due to the intractable itchiness. There have been a variety of effective methods to alter the appearance of the scar. However, the treatments for itching from hypertrophic scar are scarce. In 2009, P.Gazerani used Botox to treat histamine-induced itch with favorable results. In the clinical setting, however, the efficacy of Botox to treat itch from hypertrophic scar was yet to be proven. Therefore, the goal of this study is to conduct a randomized controlled trials about using Botox to treat itch from hypertrophic scar.

ELIGIBILITY:
Inclusion Criteria:

1. The patients undergoing laparotomy and thoracotomy in Veterans General Hospital in Kaohsiung (VGHKS) during 2003/1/1~2012/12/31
2. Hypertrophic scars containing more than two itchy sites with itchiness scale >3
3. Good wound healing condition, no infection sign
4. Age older than 20 year-old

Exclusion Criteria:

1. Allergy to Botulinum toxin
2. Inability to express self-willingness
3. Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The degree of itchiness | 6 months

SECONDARY OUTCOMES:
Pain scale | Within one minue after drug injection
  We'll ask the participant about the pain during injection. The question will be asked within one minute after drug injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Akhtar N, Brooks P. The use of botulinum toxin in the management of burns itching: preliminary results. Burns. 2012 Dec;38(8):1119-23. doi: 10.1016/j.burns.2012.05.014. Epub 2012 Jul 12. PMID 22795731
- [Background] Gazerani P, Pedersen NS, Drewes AM, Arendt-Nielsen L. Botulinum toxin type A reduces histamine-induced itch and vasomotor responses in human skin. Br J Dermatol. 2009 Oct;161(4):737-45. doi: 10.1111/j.1365-2133.2009.09305.x. Epub 2009 May 11. PMID 19624547